CLINICAL TRIAL: NCT03425656
Title: A Phase III, Randomized, Two-armed, Triple Blinded, Parallel, Active Controlled Non-Inferiority Clinical Trial of AryoTrust (AryoGen Trastuzumab) Efficacy and Safety in Comparison to Herceptin (Genentech) in HER2-Positive Breast Cancer
Brief Title: Comparing Efficacy and Safety of AryoGen Pharmed Biosimilar Trastuzumab (AryoTrust) Versus Herceptin® in Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRA.ARY.RS.95 (III)
Record Dates: First submitted 2017-11-21; First posted 2018-02-07 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-01

CONDITIONS: Malignant Neoplasm of Breast
Keywords: breast cancer; AryoTrust; Herceptin®; non-Inferiority
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab (AryoTrust) (Experimental): Trastuzumab (AryoTrust) is given concomitantly with docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide
  Interventions: Drug: Trastuzumab plus docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide
- Trastuzumab (Herceptin) (Active Comparator): Trastuzumab (Herceptin) is given concomitantly with docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide
  Interventions: Drug: Trastuzumab plus docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide

INTERVENTIONS:
Drug: Trastuzumab plus docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide — Trastuzumab (8 mg/kg IV loading dose at cycle 1, followed by 6 mg/kg at subsequent cycles) is given concomitantly with docetaxel (100 mg/m2 IV) for four 21-day cycles after four 14-day cycles of Doxorubicin (60 mg/m2 IV) plus cyclophosphamide (600 mg/m2 IV)

SUMMARY:
This is A Phase III, randomized, two-armed, patient-outcome assessor-data analyzer blinded, parallel active controlled non-Inferiority clinical trial study to evaluate efficacy and safety of AryoTrust (Aryogen Trastuzumab in comparison to Herceptin® (Genentech/Roche) in patients with Human Epidermal Growth Factor Receptor 2-Positive breast cancer. The main objective is to verify the non-inferiority of AryoTrust (Aryogen trastuzumab) vs. Herceptin® (Genentech/Roche trastuzumab), both given concomitantly with docetaxel after doxorubicin plus cyclophosphamide in the neoadjuvant setting according to pathological complete response (pCR) as primary objective and objective response (cOR), clinical complete response (cCR), clinical partial response (cPR), clinical stable disease (cSD), clinical progressive disease (cPD), breast conservation rate as Secondary objectives of this study. Evaluating the safety and immunogenicity of AryoTrust vs. Herceptin®, are also the other secondary outcomes. This study has two arms and 108 subjects will participate with a 1:1 allocation and receive mentioned treatment randomly.

DETAILED DESCRIPTION:
This is A Phase III, randomized, two-armed, patient-outcome assessor-data analyzer blinded, parallel active controlled non-Inferiority clinical trial study to evaluate efficacy and safety of AryoTrust (Aryogen Trastuzumab) in comparison to Herceptin® (Genentech/Roche) in patients with Human Epidermal Growth Factor Receptor 2-Positive breast cancer. Patients who met the following criteria will be recruited. The inclusion criteria are: 18-70 years old female patients, Patients with newly diagnosed stage III (locally advanced) or in-operable stage II (due to sizes larger than 5 cm or high tumor to breast ratio) tumors are candidates for participation, Willing and able to sign an informed consent, Pathological diagnosis of adenocarcinoma of the breast, ECOG status of 0-1, With any ER/PR status, HER2 positive (Immunohistochemical (IHC) 3+ intensity, amplification of the HER2 gene on fluorescence in situ hybridization (FISH+ ) or HER2 positive results of Chromogenic in situ hybridization (CISH)). Exclusion criteria are: Clinical or radiologic evidence of metastatic disease, History of any other malignancy including previous breast cancer, second non-breast malignant disease, History of previous chemotherapy, Left ventricular ejection fraction [LVEF] <55% confirmed by echo cardiogram within 3 months before registration, Any prior myocardial infarction, History of documented congestive heart failure (CHF),Any prior history of arrhythmia or cardiac valvular disease requiring medications or clinically significant, Current use of medications for treatment of angina pectoris, Current uncontrolled hypertension (diastolic > 100 mmHg or systolic > 200 mmHg), A severe conduction abnormality (having pacemaker or diagnosed by the ECG) and any other significant cardiovascular disease, Hematologic abnormalities including baseline Absolute Neutrophil Count (ANC) of ≤1,500/µL or platelet count ≤ 100,000/µL, Liver dysfunction including (baseline) Alanine amino transferase (ALT) and/or aspartate amino transferase (AST) ≥ 3 Upper Limit Normal (ULN), Alkaline phosphatase (ALP) ≥3 ͯ ULN, serum total, bilirubin > 1.5 ULN, Renal dysfunction, defined as serum creatinine ≥2.5 mg/dL, Pregnant, lactating women or women of childbearing potential who are not willing to use adequate contraception.

The main objective is to verify the non-inferiority of AryoTrust (Aryogen Trastuzumab) vs. Herceptin® (Genentech/Roche Trastuzumab), both given concomitantly with docetaxel after doxorubicin plus cyclophosphamide in the neoadjuvant setting according to pathological, clinical response and immunogenicity assay in patients with Human Epidermal Growth Factor Receptor 2-Positive breast cancer. The primary objective of this study is to verify the non-inferiority of AryoTrust vs. Herceptin®, given concomitantly with docetaxel after doxorubicin plus cyclophosphamide in the neoadjuvant setting according to pathological complete response (pCR) rate. The secondary objectives are to evaluate non-significance between AryoTrust and Herceptin®, given concomitantly with docetaxel after Adriamycin plus cyclophosphamide in the neoadjuvant setting according to clinical objective response (cOR), clinical complete response (cCR), clinical partial response (cPR), clinical stable disease (cSD), clinical progressive disease (cPD), breast conservation rateEvaluating the safety and immunogenicity of AryoTrust vs. Herceptin®, are also the other secondary outcomes. This study has two arms and 108 subjects will participate with a 1:1 allocation and receive AryoTrust vs. Herceptin® randomly given concomitantly with docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide For primary outcome analysis, Treatment differences in proportions will be calculated. A 95% two-sided confidence interval will be constructed and the upper bound to determine non-inferiority with a 2.5% significance level will be used.Frequency and proportions will be calculated for all secondary efficacy endpoints include clinical complete response (cCR), clinical partial response (cPR), clinical stable disease (cSD), clinical progressive disease (cPD), clinical objective response (cOR), breast conservation rate. All safety data will be analyzed descriptively by each treatment group. same protocol and procedures have been implemented by using same SOPs. Regular and strict monitoring visits have been provided to ensure all processes will be carried out in accordance with GCP. Probable variation of eligibility criteria and evaluation criteria are resolved through investigator meetings.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old female patients
* Patients with newly diagnosed stage III (locally advanced) or inoperable stage II (due to sizes larger than 5 cm or high tumor to breast ratio) tumors are candidates for participation.
* Willing and able to sign an informed consent
* Pathological diagnosis of adenocarcinoma of the breast
* ECOG status of 0-1
* With any ER/PR status
* HER2 positive (Immunohistochemical (IHC) 3+ intensity, amplification of the HER2 gene on fluorescence in situ hybridization (FISH+ ) or HER2 positive results of Chromogenic in situ hybridization (CISH+)).

Exclusion Criteria:

* Clinical or radiologic evidence of metastatic disease
* History of any other malignancy including previous breast cancer, second non-breast malignant disease
* History of previous chemotherapy
* Left ventricular ejection fraction [LVEF] <55% confirmed by echo cardiogram within 3 months before registration, Any prior myocardial infarction, History of documented congestive heart failure (CHF),Any prior history of arrhythmia or cardiac valvular disease requiring medications or clinically significant, Current use of medications for treatment of angina pectoris, Current uncontrolled hypertension (diastolic > 100 mmHg or systolic > 200 mmHg), A severe conduction abnormality (having pacemaker or diagnosed by the ECG) and any other significant cardiovascular disease.
* Hematologic abnormalities including baseline Absolute Neutrophil Count (ANC) of ≤1,500/µL or platelet count ≤ 100,000/µL
* Liver dysfunction including : (baseline)

  * Alanine amino transferase (ALT) and/or aspartate amino transferase (AST) ≥ 3 Upper Limit Normal (ULN)
  * Alkaline phosphatase (ALP) ≥3 ͯ ULN
  * serum total bilirubin > 1.5 ULN
* Renal dysfunction, defined as serum creatinine ≥2.5 mg/dL
* Pregnant, lactating women or women of childbearing potential who are not willing to use adequate contraception

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-07-09 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Safaei, M.D, Principal Investigator — Tehran University of Medical Sciences
Locations (19):
- Iran (19):
  - Shafa Hospital, Ahvāz
  - Sheikh Mofid Clinic, Isfahan
  - Javadol Aemeh Clinic, Kerman
  - Park clinic, Kerman
  - Payandeh Clinic, Kermanshah
  - Imam Reza Hospital, Mashhad
  - Tohid Hospital, Sanandaj
  - Shahid Faqihi Hospital, Shiraz
  - Baqiatallah Hospital, Tehran
  - Booali Hospital, Tehran
  - Firoozgar Hospital, Tehran
  - Imam Khomeini hospital, Tehran
  - Jahad Daneshgahi Clinic, Tehran
  - Masood Clinic, Tehran
  - Mehrad Hospital, Tehran
  - Rasool Akram Hospital, Tehran
  - Toos Hospital, Tehran
  - Mortazavizadeh Clinic, Yazd
  - Aliebne Abitaleb Hospital, Zahedan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trastuzumab (AryoTrust) | Trastuzumab (Herceptin)
Started | 54 | 54
Completed | 48 | 44
Not Completed | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab (AryoTrust) | Trastuzumab (Herceptin) | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Median (Full Range); unit: year] | 47.5 [28 to 63] | 46 [26 to 69] | 46 [26 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Median (Full Range); unit: Kg] | 70 [46 to 110] | 70 [44 to 100] | 70 [44 to 110]
Tumor Size [Median (Full Range); unit: mm] | 33 [22 to 44] | 33 [21 to 41] | 33 [21 to 44]
IHC 2+ [Number; unit: participants] — In Immunohistochemistry (IHC), different staining intensities can indicate variations in the amount or distribution of the target protein (HER2) within the tissue sample. Intensity is subjectively interpreted by an observer as "0" to "3+". IHC 2+ staining intensity suggests a moderate level of HER2 protein expression. The staining appears moderately coloured, not as dark as strong staining, but clearly observable. Staining intensity alone may not provide a complete prognosis or treatment prediction, but generally, HER2 overexpression in breast cancer is associated with poorer prognosis.
  participants | 9 | 11 | 20
IHC 3+ [Count of Participants; unit: Participants] — In Immunohistochemistry (IHC), different staining intensities can indicate variations in the amount or distribution of the target protein (HER2) within the tissue sample. Intensity is subjectively interpreted by an observer as "0" to "3+". IHC 3+ staining intensity indicates a high concentration or abundant expression of HER2 protein within the cells or tissue. It appears very dark and prominent under the microscope. Staining intensity alone may not provide a complete prognosis or treatment prediction, but generally, HER2 overexpression in breast cancer is associated with poorer prognosis.
  Participants | 45 | 43 | 88
FISH+ [Count of Participants; unit: Participants] — Herein, Fluorescence In Situ Hybridisation (FISH) involves using fluorescently labelled DNA probes that specifically bind to the HER2 gene in the tumoural cells. When these probes bind to the HER2 gene, they emit fluorescent signals that can be visualised under a fluorescence microscope. The number of signals indicates the quantity of the HER2 gene. If there are more copies (amplification) than usual, it is referred to as "FISH+". Breast cancers with HER2 gene amplification or overexpression (FISH+) tend to have more aggressive behaviour and are historically associated with a poorer prognosis.
  Participants | 3 | 2 | 5
CISH+ [Count of Participants; unit: Participants] — In this context, Chromogenic In Situ Hybridisation (CISH) involves using labelled DNA probes that bind to the HER2 gene. These probes are then visualised under a standard light microscope using chromogenic detection methods, resulting in a coloured signal that indicates the presence and quantity of the HER2 gene in the cancer cells. Indicating HER2 gene amplification or overexpression using CISH (known as CISH+) is associated with a more aggressive subtype of breast cancer with a poorer prognosis.
  Participants | 6 | 9 | 15
ER and/or PR positive [Count of Participants; unit: Participants] — The standard method for assessing oestrogen receptors (ER) and progesterone receptors (PR) status in breast cancer tissue samples is immunohistochemistry (IHC), in which tissue samples are stained with antibodies against ER and PR proteins. Then, the staining intensity and the percentage of tumour cells with positive nuclear staining are assessed. If ≥1% of tumour cells stain positive, the tumour is considered hormone receptor-positive. Among patients with HER2+ breast cancer, those with ER and/or PR typically have a better prognosis and may respond well to hormone-targeted therapies.
  Participants | 36 | 30 | 66
ER and PR negative [Count of Participants; unit: Participants] — The standard method for assessing oestrogen receptors (ER) and progesterone receptors (PR) status in breast cancer tissue samples is immunohistochemistry (IHC), in which tissue samples are stained with antibodies against ER and PR proteins. Then, the staining intensity and the percentage of tumour cells with positive nuclear staining are assessed. If <1% of tumour cells stain positive, the tumour is considered hormone receptor-negative. Among patients with HER2+ breast cancer, those without both ER and PR typically have a worse prognosis and respond less to hormone-targeted therapies.
  Participants | 18 | 24 | 42

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes
Time Frame: week 23
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab (AryoTrust) | Trastuzumab (Herceptin)
Number analyzed (Participants) | 48 | 44
Participants | 18 | 15
Statistical Analysis 1: Comparison: Trastuzumab (AryoTrust) vs Trastuzumab (Herceptin); Test type: Non-Inferiority — We used a non-inferiority margin of 0.25 for the primary endpoint; p = 0.73, Chi-squared; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.23 to 0.16]

2. Secondary Outcome: Clinical Objective Response
Description: clinical Complete Response + clinical Partial Response
Time Frame: week 21
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab (AryoTrust) | Trastuzumab (Herceptin)
Number analyzed (Participants) | 54 | 54
Participants | 41 | 35
Statistical Analysis 1: Comparison: Trastuzumab (AryoTrust) vs Trastuzumab (Herceptin); Test type: Other; p = 0.72, Fisher Exact

3. Secondary Outcome: Breast Conservation Rate
Description: Patients who underwent lumpectomy
Time Frame: week 23
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab (AryoTrust) | Trastuzumab (Herceptin)
Number analyzed (Participants) | 54 | 54
Participants | 11 | 7
Statistical Analysis 1: Comparison: Trastuzumab (AryoTrust) vs Trastuzumab (Herceptin); Test type: Other; p = 0.42, Chi-squared; Chi-squared = 0.42

4. Secondary Outcome: Safety Assessment by Evaluation of Adverse Events (AEs) and Abnormal Laboratory Results
Description: Safety assessment, including the incidence of all reported AEs and abnormal laboratory results was done. All AEs were classified based on the Medical Dictionary for Regulatory Activities (MedDRA Desktop Browser 4.0 Beta) terms as System Organ Class (SOC) and Preferred Term (PT). All the reported events were graded according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Moreover, seriousness of AEs was assessed according to International Council for Harmonization (ICH-E2B) guidelines. The causality relation was assessed based on the World Health Organization (WHO) criteria.
Time Frame: up to week 26
Population: A total of 108 patients were analyzed for AEs.Reports were based on the Safety set. The safety set included all randomized patients who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab (AryoTrust) | Trastuzumab (Herceptin)
Number analyzed (Participants) | 54 | 54
Participants | 54 | 54
Statistical Analysis 1: Comparison: Trastuzumab (AryoTrust) vs Trastuzumab (Herceptin); Test type: Non-Inferiority — We used a non-inferiority margin of 0.25 for the primary endpoint; p = 0.59, Chi-squared

5. Secondary Outcome: The Number of Participants With Anti-drug Antibodies Against Trastuzumab (AryoTrust)
Description: The levels of anti-drug antibodies against Trastuzumab ( aryotrust ) are assessed via ELISA and the percantage of positive value are reported
Time Frame: week 10, week 13, week 19, week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab (AryoTrust) | Trastuzumab (Herceptin)
Number analyzed (Participants) | 54 | 54
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion (26 weeks)
Groups:
- Trastuzumab (AryoTrust) / ACTH: Trastuzumab (AryoTrust) is given concomitantly with docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide
  Trastuzumab plus docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide: Trastuzumab (8 mg/kg IV loading dose at cycle 1, followed by 6 mg/kg at subsequent cycles) is given concomitantly with docetaxel (100 mg/m2 IV) for four 21-day cycles after four 14-day cycles of Doxorubicin (60 mg/m2 IV) plus cyclophosphamide (600 mg/m2 IV)
- Trastuzumab (Herceptin) / ACTH: Trastuzumab (Herceptin) is given concomitantly with docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide
  Trastuzumab plus docetaxel (for four 21-day cycles) after four 14-day cycles of Doxorubicin plus cyclophosphamide: Trastuzumab (8 mg/kg IV loading dose at cycle 1, followed by 6 mg/kg at subsequent cycles) is given concomitantly with docetaxel (100 mg/m2 IV) for four 21-day cycles after four 14-day cycles of Doxorubicin (60 mg/m2 IV) plus cyclophosphamide (600 mg/m2 IV)
Arm/Group | Trastuzumab (AryoTrust) / ACTH | Trastuzumab (Herceptin) / ACTH
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 42/54 | 44/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (AryoTrust) / ACTH (N=54) | Trastuzumab (Herceptin) / ACTH (N=54)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 13 | 17
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Ejection fraction decreased (Cardiac disorders) | 0 | 0
Chest pain (Cardiac disorders) | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0
Ageusia (Gastrointestinal disorders) | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0
Faecal vomiting (Gastrointestinal disorders) | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Oropharyngeal pain (Gastrointestinal disorders) | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Axillary pain (General disorders) | 0 | 0
Disease Progression (General disorders) | 0 | 0
Fatigue (General disorders) | 0 | 1
Hot flush (General disorders) | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0
Pain (General disorders) | 0 | 0
Pyrexia (General disorders) | 0 | 0
Swelling (General disorders) | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 0
Nail infection (Infections and infestations) | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 0 | 0
Hyperbilirubinaemia (Investigations) | 0 | 0
Hyperphosphataemia (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0
Headache (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0
Vertigo (Nervous system disorders) | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 44
Blister (Skin and subcutaneous tissue disorders) | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin wound (Skin and subcutaneous tissue disorders) | 1 | 0
Epistaxis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-12-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03425656/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2017-12-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03425656/SAP_001.pdf